CLINICAL TRIAL: NCT03951688
Title: Effects of a Multi-modal Exercise Program in Community-dwelling Older Adults
Brief Title: Multi-modal Exercise Program in Older Adults
Acronym: MME-CDOA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Juan F. Lisón Párraga, Dr, Head of Medicine, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: UNIVERSITY CARDENAL HERRERA-21
Record Dates: First submitted 2019-05-14; First posted 2019-05-15 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Community-dwelling Older Adults

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental-Multi-modal exercise program (Experimental): Each home-based session (48) starts with 7 minutes of moderate warm-up exercises focusing on mobility and flexibility. Secondly, the strengthening exercises consist of knee extensions, knee flexions, hip abductions, ankle plantar flexions, and ankle dorsiflexions. Thirdly, a set of balance exercises including knee bends, backwards walking, walking and turning around, sideways walking, tandem stance, tandem walk, one leg stand, heel walking, toe walking, toe to heel walking backwards, sit-to-stand, and stair walking.
  Finally, participants are instructed to walk at their usual pace for at least 10 minutes.
  Interventions: Other: Experimental-Multi-modal exercise program
- Control Group (No Intervention): No intervention

INTERVENTIONS:
Other: Experimental-Multi-modal exercise program — Each home-based session (48) starts with 7 minutes of moderate warm-up exercises focusing on mobility and flexibility. Secondly, the strengthening exercises consist of knee extensions, knee flexions, hip abductions, ankle plantar flexions, and ankle dorsiflexions. Thirdly, a set of balance exercises including knee bends, backwards walking, walking and turning around, sideways walking, tandem stance, tandem walk, one leg stand, heel walking, toe walking, toe to heel walking backwards, sit-to-stand, and stair walking.
  Finally, participants are instructed to walk at their usual pace for at least 10 minutes.
  Arms: Experimental-Multi-modal exercise program

SUMMARY:
Aim: To evaluate the short-term effects of a multi-modal exercise program on physical performance variables in older adults.

DETAILED DESCRIPTION:
* Aim: To evaluate the short-term effects of a 16 weeks home-based multi-modal exercise program on physical performance variables in community-dwelling older adults.
* Design: randomized controlled trial.
* Setting: home-based intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Community-dwelling

Exclusion Criteria:

* Unable to ambulate independently
* Mini-mental state examination score < 24
* Barthel Index score < 80
* Unstable cardiovascular disease
* Neurological disorder that could compromise exercising
* Upper or lower-extremity fracture in the past year

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2019-12-28 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Timed 'Up-and-Go' test (TUG) | 16 weeks
  The participants are instructed to stand up from a standard chair of 45 cm height, walk 3 metre, turn around a cone, return to the chair, and sit down again in the shortest time possible without running. Two trials are performed, and the quicker time in seconds is recorded. Shorter time indicates better performance.

SECONDARY OUTCOMES:
Repeated chair stand test (STS-5) | 16 weeks
  The participants are instructed to stand from a chair five successive times as quickly as possible without the assistance of their arms. Shorter time indicates better performance.
One-Leg Stand test (OLS) | 16 weeks
  Participants are instructed to start the test from a standing position with their eyes open and arms at their sides, choose a leg to stand on, flex the opposite knee, allowing the foot to clear the ground, and stand unassisted on one leg as long as possible. Longer time indicates better performance.

CONTACTS AND LOCATIONS:
Overall Officials: JF Lisón, PhD, Principal Investigator — Cardenal Herrera University
Locations (1):
- Universidad CEU Cardenal Herrera, Moncada, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided